CLINICAL TRIAL: NCT02652546
Title: A Phase 1 Study of CC-11050 in Human Immunodeficiency Virus-1-Infected Adults With Suppressed Plasma Viremia on Antiretroviral Therapy
Brief Title: CC-11050 in Human Immunodeficiency Virus-1-Infected Adults With Suppressed Plasma Viremia on Antiretroviral Therapy (APHRODITE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 160044; 16-I-0044
Record Dates: First submitted 2016-01-09; First posted 2016-01-12 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11-02

CONDITIONS: HIV, Inflammation
Keywords: HIV/AIDS; Immune Activation; Anti-Inflammatory; TNF; Phosphodieterase Inhibitor
MeSH Terms: conditions — Inflammation; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- A (Active Comparator): CC-11050 200mg (2 capsules) BID with food
  Interventions: Drug: Assess Safety; Drug: Effect of drug on viral load; Drug: Effect of drug on T-cell count; Drug: Effect of drug on inflammatory biomarkers
- B (Placebo Comparator): Placebo (2 capsules) BID with food
  Interventions: Drug: Assess Safety

INTERVENTIONS:
Drug: Assess Safety — Assess the safety of a 12-week course if CC-1150 in HIV-infected adults who have been on ART for greater than or equal to 1 year and have suppressed plasma viremia
Drug: Effect of drug on viral load — Evaluate the effect of CC-11050 on plasma HIV-1 RNA levels by both conventional and single copy assay at week 12 and over all evaluable time points
  Arms: A
Drug: Effect of drug on T-cell count — Evaluate the effect of CC-11050 on CD4+ T cell counts and percentages at week 12 and over all evaluable time points
  Arms: A
Drug: Effect of drug on inflammatory biomarkers — Evaluate the effect of CC-11050 on markers of markers of systemic inflammation (TNF, IL-^, CRP, IFNg, sCD14, D-dimer) at week 12 and over all evaluable time points.
  Arms: A

SUMMARY:
Background:

When there is a threat to the body, the immune system triggers inflammation. Too much inflammation can damage the body or cause painful symptoms. Some people with HIV feel sick after they start HIV drugs because their recovering immune systems cause too much inflammation. Or their immune systems can become activated all the time. This can cause serious health problems. Researchers want to test if the drug CC-11050 helps treat inflammation in people taking HIV drugs.

Objectives:

To test if CC-11050 is safe and well-tolerated for people with HIV who are taking HIV drugs. To see if it reduces inflammation.

Eligibility:

People ages 18 and older with HIV who have been on antiretroviral therapy for at least 1 year.

Design:

Participants will be screened with:

Medicine review

Physical exam and medical history

Blood and urine tests

Chest x-ray

Electrocardiogram (ECG): Soft electrodes on the skin record heart signals.

Participants will be randomly assigned to take capsules of either CC-11050 or a placebo. They will take the capsules every day for 12 weeks. They will continue to take their HIV drugs.

Participants will have a baseline visit within 2 months of screening. This includes:

Physical exam and medical history

Blood and urine tests

ECG

Leukapheresis: Blood is removed by a needle in one arm and passed through a machine that removes white blood cells. The rest of the blood is returned through a needle in the other arm.

Participants will have follow-up visits 2, 4, 8, 12, and 16 weeks after the baseline visit. These may include repeats of some of the baseline tests.

DETAILED DESCRIPTION:
CC-11050 is a novel anti-inflammatory compound with potential to treat a variety of chronic inflammatory conditions and cytokine storms associated with infectious diseases. CC-11050 is a selective phosphodiesterase-4 inhibitor (PDE4) that is active in several in vivo models of inflammatory disease, inhibiting systemic TNF- production, colitis symptoms of the colon, psoriasiform features in the skin, arthritogenic swelling in the joints, neutrophilia and eosinophilia in the lung, and reducing choroidal neovascularization. These data suggest that CC-11050 may have therapeutic potential for chronic inflammatory conditions and/or as an antiangiogenic treatment. The safety profile of CC-11050 has been investigated in healthy males and in subjects with cutaneous lupus erythematosus; the most frequently reported adverse events were fatigue, headache, upper respiratory infection and pruritus; there were no deaths or serious adverse events.

Inflammation is an important contributor to HIV pathogenesis both prior to and after ART initiation. Inflammatory responses can occur abruptly upon ART initiation (known as immune reconstitution inflammatory syndrome or IRIS) and can be chronic in persons with suppressed plasma HIV viremia who are treated with ART, and has been linked to an excess risk of non-AIDS serious events such as cardiovascular, liver and kidney disease and accelerated bone loss. Corticosteroids to reduce levels of inflammatory cytokines in plasma are a standard therapeutic intervention for IRIS, however a more targeted anti-inflammatory and less broadly immunosuppressive intervention is desirable.

We propose a double-blind, randomized trial to assess the safety of CC-11050 in adults with HIV infection who have taken ART for at least 1 year and have suppressed plasma viremia. Enrolled subjects will be randomized 2:1 to 200 mg CC-11050 or placebo twice daily for 12 weeks. Participants will be evaluated at weeks 0, 2, 4, 8, 12 and 16. Changes in in plasma HIV-1 RNA levels (by clinical assay), CD4+ T cell counts and percentages, and the effect on markers of systemic inflammation (e.g., TNF, IL-6, CRP, IFNg, sCD14, D-dimer) will be measured. The effect of CC-11050 on cellular immune activation (T cells and monocytes), and on viral reservoirs (cell associated HIV DNA and RNA) will also be assessed.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adults (greater than or equal to 18 years)
  2. Body mass index (BMI) less than or equal to 35 kg/m2
  3. On ART for a minimum of 1 year and on a stable regimen (according to DHHS guidelines) for at least 3 months prior to screening
  4. Plasma HIV-1 RNA level <50 copies/mL at screening (patients with 50-499 <500 copies/mL at screening may be asked to return for rescreening in four (4) weeks or later
  5. Men and women must be willing to take appropriate precautions to prevent pregnancy as described below
  6. Willingness to undergo genetic testing
  7. Willingness to allow storage of specimens for future analysis
  8. Negative serum or urine pregnancy test (for women of childbearing potential)
  9. Under the care of a primary care physician outside of the NIH

Contraception: The effects of CC-11050 on the developing human fetus are unknown. For this reason, subjects must agree to not become pregnant. Females of childbearing potential must have a pregnancy test before initiating the study agent and at each study visit. Because of the risk involved, male and female study participants who engage in sexual activities that can result in pregnancy must agree to use of a male or female condom at every potentially reproductive sexual encounter, AS WELL AS one of the other methods listed below, beginning at the baseline visit and continuing until 3 months after discontinuation of the study agent. Acceptable methods are as follows:

* Hormonal contraception [e.g. consistent use of oral contraceptive pill daily or other hormonal method such as contraceptive implant or injection] (must be started 1 month prior to receiving the first dose of study agent)
* Diaphragm or cervical cap
* Intrauterine device (IUD)
* Male partner with a vasectomy

During the study, if a participant becomes pregnant or suspects they are pregnant, they should inform the study staff and their primary care physician immediately. The study medication will be stopped immediately and if on CC-11050 they will be referred to a high risk pregnancy specialist and followed by the study team for the remainder of the pregnancy or the rest of the study, whichever occurs later.

EXCLUSION CRITERIA:

1. Body mass index (BMI) less than or equal to 18.5 kg/m2
2. Protease inhibitor-based ART regimen
3. ART regimen which includes Cobicistat
4. Absence of alternate available ART options in case of virologic failure
5. Serum ALT or AST value Grade >2 or total bilirubin greater than the ULN unless it is indirect due to Gilbert s disease
6. History of chronic hepatitis B (+HbsAg or +HBV DNA in plasma) and/or C - treated chronic hepatitis C with SVR > 2 years will be accepted.
7. Cirrhosis of the liver, or any known active or chronic liver disease
8. Recent history (<30 days) of infection requiring inpatient hospitalization or systemic therapy
9. Depression. Patients who report depression or, are suspected or known to have depression and are on stable anti-depressants will undergo Psychiatry evaluation and clinical assessments to determine eligibility. These assesments will be done by a psychiatrist and may include: Beck Depression Inventory (BDI), Spielberger State-Trait Anxiety Inventory (STAI), Montreal Cognitive Assessment(MoCA). The BDI, STAI, and MoCA will be administered to patients being considered for study enrollment. The BDI and STAI may be repeated at least once during follow-up visits in those deemed eligible to participate.
10. Current breastfeeding
11. Current or anticipated treatment with immunomodulating agents (such as systemic corticosteroids, interleukins, interferons) or any agent with known anti-HIV activity (other than antiretrovirals approved for use in the treatment of HIV)
12. Any experimental medications within 4 weeks prior to screening or anticipated use of such medications during the trial.
13. Current (4 weeks prior to the first dose of study drug,) or anticipated use of antimetabolites; alkylating agents; or drugs other than ART, herbal preparations (including St. John s wort), and foods (including grapefruit) known to affect activity of the CYP3A4 enzyme pathway
14. Use of thalidomide, lenalidomide, pomalidomide, systemic corticosteroids within 4 weeks of screening
15. Any prior history of PDE4 inhibitor use
16. History of pancreatitis, elevated lipase (less than or equal to 1.5 above the upper limit of normal) or triglyceride level >500 mg/dL.
17. History of clinically significant metabolic, endocrine, hepatic, renal, hematologic, pulmonary, gastrointestinal, autoimmune or cardiovascular disorders
18. Uncontrolled hypertension (persistent measurements over 140/90)
19. Bradycardia, defined as a sinus rhythm <50 beats/min (bpm)
20. History or presence of a clinically significant abnormal ECG
21. History of malignancy except cured basal or squamous cell carcinoma of the skin or cutaneous Kaposi s sarcoma not requiring systemic therapy during the trial
22. Receipt of radiation or cytotoxic chemotherapeutic agents, unless fully recovered from disease by the time of the first dose of study drug as determined by the opinion of the Investigator, or anticipated use of such agents during the study period
23. Any condition or significant problems that, based on the judgment of the investigator, would increase risk to the subject or would interfere with the subject s ability to comply with protocol requirements.

Co-enrollment Guidelines: Co-enrollment in other trials is restricted, other than enrollment on observational studies or those evaluating the use of a licensed medication. Study staff should be notified of co-enrollment as it may require the approval of the study investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-01-09; Primary Completion 2017-05-15 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of AEs and SAEs in subjects receiving study agent vs placebo | 12/30/2016

SECONDARY OUTCOMES:
Plasma HIV-1 RNA levels by both conventional and single-copy assay at Weeks 0,2,4,8, and 12 | week 12
CD4+ T cell counts and percentages at weeks 2,4,8 and 12 | week 12
Markers of systemic inflammation (TNF, IL-6, CRP, IFNy, sCD14, D-dimer) at weeks 2,4,8 and 12 | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Irini Sereti, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Andrade BB, Singh A, Narendran G, Schechter ME, Nayak K, Subramanian S, Anbalagan S, Jensen SM, Porter BO, Antonelli LR, Wilkinson KA, Wilkinson RJ, Meintjes G, van der Plas H, Follmann D, Barber DL, Swaminathan S, Sher A, Sereti I. Mycobacterial antigen driven activation of CD14++CD16- monocytes is a predictor of tuberculosis-associated immune reconstitution inflammatory syndrome. PLoS Pathog. 2014 Oct 2;10(10):e1004433. doi: 10.1371/journal.ppat.1004433. eCollection 2014 Oct. PMID 25275318
- [Background] Schafer PH, Chen P, Fang L, Wang A, Chopra R. The pharmacodynamic impact of apremilast, an oral phosphodiesterase 4 inhibitor, on circulating levels of inflammatory biomarkers in patients with psoriatic arthritis: substudy results from a phase III, randomized, placebo-controlled trial (PALACE 1). J Immunol Res. 2015;2015:906349. doi: 10.1155/2015/906349. Epub 2015 Apr 20. PMID 25973439
- [Background] Marzi A, Feldmann H. Ebola virus vaccines: an overview of current approaches. Expert Rev Vaccines. 2014 Apr;13(4):521-31. doi: 10.1586/14760584.2014.885841. Epub 2014 Feb 27. PMID 24575870